CLINICAL TRIAL: NCT06099873
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Trial of ZX-7101A Tablets to Evaluate the Efficacy and Safety in the Treatment of Uncomplicated Influenza in Adolescents
Brief Title: Study to Assess the Safety and Efficacy of ZX-7101A in Adolescents With Influenza
Acronym: ZX-7101A-207
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZX-7101A-207
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Viral Infection
Keywords: adolescent; ZX-7101A

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, placebo-controlled Phase III clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZX-7101A (Experimental): Before starting study treatment on day 1 (D1), eligible subjects were randomly assigned in a 1:1 ratio to receive either ZX-7101A (1 tablet，specification：40mg, single dose) or placebo (1 tablet, single dose).
  A total of 360 subjects were planned to be enrolled in this study，in ZX-7101A group was planned to enroll about 180 subjects.
  Interventions: Drug: ZX-7101A
- Placebo group (Placebo Comparator): Before starting study treatment on day 1 (D1), eligible subjects were randomly assigned in a 1:1 ratio to receive either ZX-7101A (1 tablet，specification：40mg, single dose) or placebo (1 tablet, single dose).
  A total of 360 subjects were planned to be enrolled in this study，in placebo group was planned to enroll about 180 subjects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZX-7101A — Day1 Take one tablet of ZX-7101A orally once (specification: 40mg/ tablet) with appropriate amount of warm water
  Arms: ZX-7101A
Drug: Placebo — Day1 Take one tablet of Placebo orally once with appropriate amount of warm water
  Arms: Placebo group

SUMMARY:
The primary object of this study is evaluating the efficacy of ZX-7101A tablets versus placebo in the treatment of uncomplicated simple influenza in adolescents.

The seongdary object is evaluating the safety of ZX-7101A tablet in the treatment of uncomplicated simple influenza in adolescents.

DETAILED DESCRIPTION:
In this study, adolescents aged 12 and < 18 with uncomplicated influenza are selected as subjects. Typical systemic and/or respiratory influenza symptoms were required, and the time interval between the first onset of influenza symptoms and random enrollment was less than 48 hours. This study is divided into screening/treatment period (D1) and observation period (about 2 weeks). You will be eligible before starting study therapy on day 1 (D1). Participants were randomly assigned 1:1 to ZX-7101A group (dose 40 mg, administration once) or placebo group (dose 1 placebo tablet, administration once), with 180 participants planned to be included in each group, for a total of about 360 participants.

ELIGIBILITY:
Inclusion Criteria:

1.≥12 to<18 years of age at the time of randomization, males or females. 2.Patients in the screening period met the following criteria:

1. Rapid influenza diagnostic test (RIDT) or polymerase chain reaction (PCR) test positive;
2. Axillary temperature ≥ 37.5℃ at screening; If taking antipyretics, axillary temperature ≥ 37.5℃ after taking the drug (more than 4 hours).
3. At least one of influenza -related systemic symptoms is moderate or greater in severity: a. muscle or joint pain, b. fatigue, c. headache, d. fever.
4. At least one of the influenza-related respiratory symptoms is moderate or greater in severity: a. nasal congestion, b. sore throat, c. cough.

3.The first occurrence of influenza symptoms ≤ 48 hours from the time of patient randomization.

1. Body temperature ≥ 37.5 ℃ (axillary temperature) or 37.5 ℃ (oral temperature) or 38.0 ℃ (rectal or tympanic membrane temperature)for the first time;
2. Or at least one systemic or respiratory symptom may occur: a. nasal congestion, b. sore throat, c. cough, d. muscle or joint pain, e. fatigue, f. headache, g. fever.

4.Be able to comply with all the study procedures, complete the subject diary as required(The guardian is allowed to fill in if necessary).

5.The subject and his/her guardian are volunteer to participate in the study and sign the written informed consent form (ICF).

6.The subject agree to maintain abstinence or take reliable contraceptive methods during the trial and persist in until 3 months after the administration of the investigational product.

Exclusion Criteria:

1. Patients with severe influenza virus infection requiring inpatient treatment.(Meet any one of the following criteria) （1）Severe cases with one of the following conditions： Persistent high fever for more than 3 days, accompanied by severe cough, purulent sputum, bloody sputum, or chest pain; Fast breathing rate, difficulty breathing, cyanosis of lips; Delayed response, drowsiness, restlessness, and other mental changes or seizures; Severe vomiting, diarrhea, and dehydration symptoms; Concomitant pneumonia; Significant exacerbation of existing underlying diseases; Other clinical situations that require hospitalization. （2）Critical cases with one of the following conditions(Including but not limited to)： Respiratory failure; Acute necrotizing encephalopathy; Shock; Multiple organ dysfunction; Other serious clinical situations that require monitoring and treatment.
2. High risk population for severe cases. (Meet any one of the following criteria):

（1）Accompanied by the following basic diseases and judged by the investigators to be clinically significant, such as lung diseases, liver diseases, kidney diseases, hematological system diseases, heart diseases, neurological and neuromuscular diseases that affect the ability to clear respiratory secretions, metabolic and endocrine system diseases, etc; （2）Subjects with low immune function, such as malignant tumors, organ or bone marrow transplants, HIV infections, or those who have been taking immunosuppressants for the past 3 months; （3）Clinical significance of correcting QT interval abnormalities in electrocardiogram display; (QTc>440ms in male or QTc>450ms in female); （4）Subjects who require long-term use of drugs containing aspirin or salicylates : It is necessary to take medication containing aspirin or salicylate regularly every day for more than 14 days; （5）BMI exceeds the standards. 3.Bronchitis, pneumonia, pleural effusion or interstitial disease confirmed by chest imaging [X-ray (anteroposterior or anteroposterior)/CT] and judged clinically significant by the investigator at screening.

4.Subjects who have developed acute respiratory tract infection, otitis media, and sinusitis within 2 weeks before screening.

5.Subjects with other infections requiring systemic anti-infective treatment, or blood routine examination at screening: <13 years of age ：white blood cell count (WBC) > 11.3 × 109/L(venous blood);≥13 to<18 years of age ：white blood cell count (WBC) > 11.0 × 109/L(venous blood).

6.Subjects with purulent sputum or suppurative tonsillitis. 7.Have difficulty in swallowing drugs or have a history of gastrointestinal diseases that seriously affect drug absorption.

8.Suspected allergic to active ingredients or excipients of the investigational product.

9.Body weight < 20 kg. 10.Medications against influenza virus within 7 days before screening. 11.Have received live vaccines or attenuated live vaccines within 14 days before randomization, influenza vaccines within 6 months before randomization.

12.Suspected or confirmed a history of alcohol or drug abuse.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 361 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
The time to the remission of all influenza symptoms (hours) | From accepting ZX-7101A until the 15 days after the first dosing
  Defined as the time from the start of study treatment to the time all flu symptoms are relieved. Symptom relief was defined as all seven influenza symptoms assessed by the subject on the subject diary card(Stuffy nose, sore throat, cough, muscle or joint pain, fatigue, headache, fever or chills/sweating) were 0 (asymptomatic) or 1 (mild)，nd the duration is at least 21.5 hours (approximately 24 hours -10%)

SECONDARY OUTCOMES:
The time influenza RNA turns negative | From accepting ZX-7101A until the 15 days after the first dosing
  Defined as the time from initiation of treatment until the first influenza viral RNA falls below the lower limit of quantification (measured by RT-PCR)
The time Virus Titer turns negative | From accepting ZX-7101A until the 15 days after the first dosing
  Defined as the time from initiation of treatment until the first viral titer falls below the lower limit of quantification
Percentage of subjects with RT-PCR positive influenza virus RNA and measurable virus titer at each visit (unit: %) | From accepting ZX-7101A until the 15 days after the first dosing
  the number of subjects with RT-PCR positive influenza virus RNA and measurable virus titer /The number of subjects
Time (in hours) for relief of 4 systemic symptoms (muscle or joint pain, weakness, headache, fever, or chills/sweating) | From accepting ZX-7101A until the 15 days after the first dosing
  Symptom remission is defined as a score of 0 (asymptomatic) or 1 (mild) for all four of the above symptoms. The duration is at least 21.5 hours
  (About 24 hours -10%)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University affiliated Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The results of the trial will be used for New Drug Application.